CLINICAL TRIAL: NCT06596733
Title: Clinical Investigation to Evaluate the Efficacy and Safety of Vit-A-Vision® When Used in Dry Eye Disease
Brief Title: Vit-A-Vision® Clinical Investigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OmniVision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vit-A-2023
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Burning Eye; Irritation; Eyeball; Tired Eye; Dry Eye Disease
MeSH Terms: conditions — Eye Burns; Asthenopia; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vit-A-Vision (Experimental): Application of Vit-A-Vision ointment
  Interventions: Device: Vit-A-Vision

INTERVENTIONS:
Device: Vit-A-Vision — Participants will apply Vit-A-Vision ointment on a daily basis, up to 3 times daily per eye, for at least 30 days.

SUMMARY:
Symptoms of ocular discomfort include dryness, burning, stinging, photophobia, foreign body sensation and contact lens intolerance. These symptoms may affect basic daily activities, such as reading, driving, and working with computers. In case of moderate to severe conditions, dry eye disease is also associated with significant pain. Dry eye disease (DED) affects hundreds of millions of people throughout the world and is one of the most frequent causes of patient visits to eye care practitioners. Diagnosing, staging and determining the efficacy of therapy in DED is often challenging due to low correlation between signs and symptoms. Furthermore, its management is complicated because of its multifactorial aetiology. In general, management approaches begin with conventional, low-risk and easily accessible patient-applied therapies such as over-the-counter lubricants for early-stage disease, and progress to more advanced therapies for more severe forms of DED. In this regard, tear supplementation with ocular lubricants (artificial tears) is considered the first-line therapy and is often the only therapy used in mild to moderate disease. They are used in all stages of dry eye, either alone (in mild to moderate disease) or in combination with other treatments (in moderate to severe disease). Most tear supplements act as lubricants. Other actions may include replacement of deficient tear constituents, dilution of proinflammatory substances, reduction of tear osmolarity and protection against osmotic stress. A wide variety of artificial tear products is currently available. These products differ with respect to several variables, that include electrolyte composition, osmolarity/osmolality, viscosity, the presence or absence of preservatives and the presence or absence of compatible solutes. Although they are all considered as standard of care in treatment of dry eye disease, the effects of many of the available products have not been evaluated in clinical investigations.

Vit-A-Vision is an ointment for ophthalmic application that relieves symptoms such as burning, irritation, slight irritation, dryness or tiredness of the eyes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Ocular Surface Disease Index (OSDI) ≧ 16
* Median of three consecutive non-invasive tear film break-up time (NIBUT) test results less than or equal to 10 seconds in at least one eye
* Willingness to apply the medical device under evaluation as per Instructions for Use (IfU) during the entire study duration (i.e., 33 ± 3 days)
* Willingness to undergo a follow-up visit at day 15 ± 3 and 33 ± 3 after enrolment
* Good understanding of written and oral speaking languages used at the centre where the study will be carried out

Exclusion Criteria:

* Known hypersensitivity (allergy) to any of the ingredients of Vit-A-Vision: vaseline, paraffin, adeps lanae, vitamin A palmitate, dexpanthenol, α-Tocopherol acetate or cetylstearyl alcohol.
* Severe forms of dry eye syndrome with OSDI > 55
* Not willing to discontinue contact lens use during the study period
* Refractive surgery within the last 12 months and/or any other ocular surgery or ocular trauma/injury within the last 4 months
* Acute inflammatory or ocular surface disease, Sjögren's Syndrome (autoimmune disease), Stevens-Johnson Syndrome, ocular pemphigoid, and radiation-induced dry eye.
* Use of systemic medication that could affect vision or dry eye, including essential fatty acids, unless dose has been constant for more than 3 months and is not expected to change during the study
* Systemic concomitant medications:

  * Corticosteroids within 2 months before enrolment and for the whole study period and / or
  * Tetracyclines within 1 month before selection and for the whole study period.
  * Vitamin A supplements intake
* Use of topical ophthalmic medication during the study or within 2 weeks prior to the first visit, other than artificial tears
* Use of topical cyclosporine within 3 months prior to the first visit
* Use of other eye drops/sprays (based on liposomic and/or oily products) during the present investigation
* Abnormality of the nasolacrimal drainage apparatus
* Permanent occlusion of lacrimal puncta in any eye
* Use of temporary punctal plug in any eye within 2 months before the selection visit
* Previous enrolment into the current investigation
* Patients who participated in any other clinical trial within the last 30 days before selection
* Children, pregnant and breastfeeding women
* Participants under the influence of excessive alcohol, narcotics or benzodiazepines
* Other diseases or characteristics judged by the investigator to be incompatible with the frequent assessments needed in this study or with reliable instillation of the products (for example: mental or physical incapacity, language comprehension, psychological disorders, dementia, geographical localisation, etc...).
* Individuals who are deprived of liberty pursuant to an administrative order or court order or approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Performance - NIBUT | After 30 days of treatment
  Improvements of the Non-Invasive tear film Break Up Time (NIBUT) after 30 days treatment with Vit-A-Vision in comparison to baseline measurements. The NIBUT measurement is an objective measure in seconds, carried out performing a test using a slit lamp.
Primary Performance - OSDI | After 30 days of treatment
  Improvements of the Ocular Surface Disease Index (OSDI) after 30 days treatment with Vit-A-Vision in comparison to baseline measurements. The OSDI is calculated using a 12-item questionnaire assessing the frequency of symptoms, environmental triggers and vision related quality of life. The score ranges from 0 (best) to 100 (worst).

SECONDARY OUTCOMES:
Secondary Performance - DEQ-5 & symptoms questionnaire | After 30 days of treatment
  Improvements of the five item Dry Eye Questionnaire (DEQ-5) and symptoms questionnaire after 30 days treatment with Vit-A-Vision in comparison to baseline measurements. The DEQ-5 is a 5 questions questionnaire assessing watery eye, discomfort, dryness, late day discomfort and dryness intensity. The maximum (worst) score is 22. A symptoms questionnaire was added to complement the DEQ-5.
Secondary Performance - ocular surface staining | After 30 days of treatment
  Improvements of the ocular surface staining with fluorescein after 30 days treatment with Vit-A-Vision, in comparison to baseline measurements. Conjunctival staining will be graded according to the TFOS (Tear Film and Ocular Surface Society) staining pattern on cornea (5 fields) and conjunctiva (4 field quadrants) using an ocular staining score from 0 (no dots) to 3 (completely spotted).
Secondary Performance - Conjunctival bulbar redness | After 30 days of treatment
  Improvements of the conjunctival bulbar redness after 30 days treatment with Vit-A-Vision, in comparison to baseline measurements. Conjunctival bulbar redness data will be collected from photographs, comparing the ones taken before and after use of device and it will be graded with 0 for no difference, 1 for more red, and 2 for less red.
Secondary Performance - Schirmer test | After 30 days of treatment
  Improvements of the Schirmer test after 30 days treatment with Vit-A-Vision, in comparison to baseline measurements. The Schirmer test provides an estimation of stimulated reflex tear flow and the normal range is ≧ 10 mm, with lower values corresponding to more severe dry eye disease.

OTHER OUTCOMES:
Safety - Adverse Events | During the study period (up to 30 days)
  Safety of the device will be assessed by systematically reporting any device or procedure related adverse events and serious adverse events (description, severity, relation to the procedure) and by monitoring the frequency and incidence of these events.
Safety - Device Deficiencies | During the study period (up to 30 days)
  Safety of the device will be assessed by systematically reporting device deficiencies (description of the deficiency) and by monitoring the frequency and incidence of these events
Acceptability | After 30 days of treatment
  Subjective end-user experience after 30 days treatment with Vit-A-Vision using a questionnaire for evaluation of product acceptance and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Schrage, Prof. Dr., Principal Investigator — Dept. of Ophthalmology Cologne Merheim
Locations (1):
- Dept. of Ophthalmology Cologne Merheim, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No